CLINICAL TRIAL: NCT05585060
Title: The Relevance and Consistency Study of Changes in End Expiratory Lung Impedence Measured by EIT and End Expiratory Lung Volume Measured by Passive Expiratory in Controlled Mechanical Ventilated Exacerbation COPD Patients
Brief Title: The Changes in End Expiratory Lung Impedence Measured by EIT and End Expiratory Lung Volume Measured by Passive Expiratory in Controlled Mechanical Ventilated Exacerbation COPD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, FuWei, Principal Investigator, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FAHGuangzhou_20220711
Record Dates: First submitted 2022-10-15; First posted 2022-10-18 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: COPD
Keywords: COPD; dynamic pulmonary hyperinflation; mechanical ventilation; end expiratory lung impedence
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEEP titration for mechanical ventilated AECOPD patients (Experimental): Pre- and post-self-controlled trials for invasive mechanical ventilated AECOPD patients during PEEP titration.
  Interventions: Diagnostic Test: the changes of end expiratory lung impedence; Diagnostic Test: the changes of end expiratory lung volume

INTERVENTIONS:
Diagnostic Test: the changes of end expiratory lung impedence — the changes of end expiratory lung impedence measured by EIT
  Other Names: △EELI
Diagnostic Test: the changes of end expiratory lung volume — the changes of end expiratory lung volume measured by apnea method
  Other Names: △EELV

SUMMARY:
The pathophysiological characteristics of respiratory failure on exacerbation of chronic pulmonary obstructive disease are the rapid deteriorate of respiratory symptoms, combined with aggravated flow limitation, gas trapping, dynamic pulmonary hyperinflation (DPH), therefore the intrinsic PEEP (PEEPi) increases. It is worthwhile to explore bedside methods to quantify the changes in dynamic pulmonary hyperinflation to guide safe and effective mechanical ventilation in airflow limited patients.

DETAILED DESCRIPTION:
The study hypothesizes that the electrical impedence tomography (EIT) measured the changes of end expiratory lung impedence (△EELI） could accurately predict the changes of end expiratory lung volume （△EELV） measured by passive expiratory in controlled mechanical ventilated exacerbation COPD patients. The research intended to conduct a research to explore the relationship between △EELI and △EELV induced by external PEEP changes in ventilated exacerbation COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* 2022.7-2023.1 exacerbation COPD invasive ventilated patients admitted to the first affiliated Guangzhou medical university; 35 to 80 years old; in stable condition judged by clinicians

Exclusion Criteria:

* SpO2<88%; instable hemodynamic (MAP<65mmHg；Norepinephrine> 0.1ug/kg.min); pregnancy; 4 hour intravenous diuretics use before research; chest deformity and trauma, subpleural pulmonary bulla; implanted electronic devices(cardiac pacemaker, implantable cardioversion defibrillator,ect); tumour or other organ dysfunction; refuse to signature the informed consent

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2023-10-08 (Estimated); Study Completion 2023-10-08 (Estimated)

PRIMARY OUTCOMES:
the changes of end expiratory lung volume | 10 minutes
  measured by EIT and IC maneuver

SECONDARY OUTCOMES:
intrinsic PEEP | 10 minutes
  measured by Esophageal balloon catheters

CONTACTS AND LOCATIONS:
Overall Officials: Rongchang Chen, PhD, Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No